CLINICAL TRIAL: NCT03299582
Title: PREventing CHemotherapy Induced Neuropathy (PreChIN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2013/00343
Record Dates: First submitted 2017-09-11; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN)
Keywords: paclitaxel; neuropathy; hypothermia; cryocompression
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: The first part of this study is in healthy subjects, followed by breast cancer patients receiving paclitaxel to study the effect of limb hypothermia in the prevention of chemotherapy-induced neuropathy.
  The second part of this study is to study the effect of cryocompression in the prevention of chemotherapy-induced neuropathy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy subjects (Hypothermia) (Experimental): To investigate the safety and tolerability of limb hypothermia in subjects without cancer
  Interventions: Device: Hypothermia
- Healthy subjects (Cryocompresion) (Experimental): To investigate the safety and tolerability of cryocompression in subjects without cancer
  Interventions: Device: Cryocompression
- Cancer subjects (Hypothermia) (Experimental): To investigate the safety and tolerability of limb hypothermia in subjects with breast cancer being treated with paclitaxel chemotherapy.
  Interventions: Device: Hypothermia
- Cancer subjects (Cryocompresion) (Experimental): To investigate the safety and tolerability of cryocompression in subjects with cancer being treated with taxane-based chemotherapy.
  Interventions: Device: Cryocompression

INTERVENTIONS:
Device: Hypothermia — Healthy subjects will undergo 3 hours of hypothermia at various temperature levels.Cancer subjects will undergo 4 hours of hypothermia during every cycle of chemotherapy.
  Arms: Cancer subjects (Hypothermia); Healthy subjects (Hypothermia)
Device: Cryocompression — Healthy subjects will undergo 3 hours of cryocompression. Cancer subjects will undergo a minimum duration of 2 hours and a maximum duration of up to 4 hours of cryocompression during every cycle of chemotherapy.
  Arms: Cancer subjects (Cryocompresion); Healthy subjects (Cryocompresion)

SUMMARY:
The project is designed to study the use of localized hypothermia alone, or with compression to the limbs during chemotherapy infusion for the prevention of chemotherapy induced peripheral neuropathy (CIPN). As a pilot study, safety, tolerability and early clinical activity will be studied. The study will be conducted on healthy volunteers and cancer patients receiving taxane chemotherapy.

DETAILED DESCRIPTION:
Localized limb hypothermia during chemotherapeutic infusion may prevent a common side effect of chemotherapy: chemotherapy-induced peripheral neuropathy (CIPN). There are no reliable methods for the prevention or the treatment of CIPN. On the basis of the dose-related pathophysiology of CIPN, the investigators hypothesize that reducing the delivery of the toxic chemotherapeutic agents to the peripheral nerves by reducing blood flow through hypothermia may reduce the occurrence of CIPN. The proposed potential treatment method would aim to reduce the development of CIPN. This project comprises of a healthy subject trial to investigate the best tolerated temperature which will be used in cancer subject trial to investigate the safety and tolerability of hypothermia or cryocompression (hypothermia with pressure) in the prevention of CIPN in cancer subjects undergoing taxane-based chemotherapy.

ELIGIBILITY:
The inclusion criterion for the healthy subjects

* Age 21-80 years
* Signed informed consent from patient
* No history of neuropathy
* ECOG 0
* No history of hospitalization in the past 6 months

The inclusion criteria for the cancer patients undergoing taxane-based chemotherapy

* Age 21- 80 years.
* Signed informed consent from patient or legal representative.
* Scheduled to receive taxane-based chemotherapy

The exclusion criteria for both healthy subjects and cancer patients

* Open skin wound or ulcers of the limbs
* A score of more than 5 in the Total Neuropathy Score (TNS) at baseline (Not applicable for healthy subjects)
* History of Raynaud's phenomenon, peripheral vascular disease, or poorly controlled diabetes

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Number of healthy subjects with treatment-related intolerance as assessed by CTCAE v4.0 and tolerability scales undergoing limb hypothermia or cryocompression | From the start of assessment until study completion, an average of 3 years
Number of cancer patients with treatment-related intolerance as assessed by CTCAE v4.0 and tolerability scales undergoing limb hypothermia or cryocompression | From the start of assessment until study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Chan, Principal Investigator — National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomchuk D, Rubley MD, Holcomb WR, Guadagnoli M, Tarno JM. The magnitude of tissue cooling during cryotherapy with varied types of compression. J Athl Train. 2010 May-Jun;45(3):230-7. doi: 10.4085/1062-6050-45.3.230. PMID 20446835
- [Background] Murgier J, Cassard X. Cryotherapy with dynamic intermittent compression for analgesia after anterior cruciate ligament reconstruction. Preliminary study. Orthop Traumatol Surg Res. 2014 May;100(3):309-12. doi: 10.1016/j.otsr.2013.12.019. Epub 2014 Mar 25. PMID 24679367